CLINICAL TRIAL: NCT01192776
Title: Optimizing Cooling Strategies at < 6 Hours of Age for Neonatal Hypoxic-Ischemic Encephalopathy
Brief Title: Optimizing (Longer, Deeper) Cooling for Neonatal Hypoxic-Ischemic Encephalopathy(HIE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial closed for emerging safety profile and futility analysis and will not resume.
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0043; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024139 (NIH); UL1RR024979 (NIH); UL1RR025008 (NIH); UL1RR025744 (NIH); UL1RR025747 (NIH); UL1RR025761 (NIH); UL1RR025764 (NIH); U10HD068284 (NIH); U10HD068278 (NIH); U10HD068270 (NIH); U10HD068263 (NIH); U10HD068244 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-06

CONDITIONS: Infant, Newborn; Hypoxia, Brain; Hypoxia-Ischemia, Brain; Encephalopathy, Hypoxic-Ischemic; Hypoxic-Ischemic Encephalopathy; Ischemic-Hypoxic Encephalopathy
Keywords: NICHD Neonatal Research Network; Hypoxic-ischemic encephalopathy (HIE); Hypothermia; Neonatal depression; Perinatal asphyxia; Fetal acidosis
MeSH Terms: conditions — Hypoxia, Brain; Hypoxia-Ischemia, Brain; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 33.5°C for 72 hours (Active Comparator): Target Temp: 33.5°C Duration: 72 hrs
  Interventions: Procedure: Whole-body Cooling
- 33.5°C for 120 hours (Experimental): Target Temp: 33.5°C Duration: 120 hrs
  Interventions: Procedure: Whole-body Cooling
- 32.0°C for 72 hours (Experimental): Target Temp: 32.0°C Duration: 72 hrs
  Interventions: Procedure: Whole-body Cooling
- 32.0°C for 120 hours (Experimental): Target Temp: 32.0°C Duration:120 hrs
  Interventions: Procedure: Whole-body Cooling

INTERVENTIONS:
Procedure: Whole-body Cooling — Whole-body cooling using a Blanketrol II or III to reach either a target core temperature of 33.5°C or 32.0°C for a duration of either 72 hours or 120 hours.
  Other Names: Blanketrol II Model 222R; Blanketrol III Model 233 (used in the II mode)

SUMMARY:
The Optimizing Cooling trial will compare four whole-body cooling treatments for infants born at 36 weeks gestational age or later with hypoxic-ischemic encephalopathy: (1) cooling for 72 hours to 33.5°C; (2) cooling for 120 hours to 33.5°C; (3) cooling for 72 hours to 32.0°C; and (4) cooling for 120 hours to 32.0°C. The objective of this study is to evaluate whether whole-body cooling initiated at less than 6 hours of age and continued for 120 hours and/or a depth at 32.0°C in will reduce death and disability at 18-22 months corrected age.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a rare, but life-threatening condition characterized by brain injury due to asphyxia diagnosed at or shortly after birth. According to the World Health Organization, more than 722,000 children died from birth asphyxia and birth trauma worldwide in 2004. An estimated 50-75 percent of infants with severe (stage 3) HIE will die, with 55 percent of these deaths occurring in the first month. Up to 80 percent of infants who survive stage 3 HIE develop significant long-term disabilities, including intellectual disabilities, epilepsy, and cerebral palsy with hemiplegia, paraplegia, or quadriplegia; 10-20 percent develop moderately serious disabilities; and up to 10 percent are normal.

Previous studies have shown treatment with hypothermia to be an effective therapy for HIE. Currently, infants diagnosed with HIE at less than six hours of age are given whole-body cooling, decreasing their core body temperature to 33.5°C (93.2° Fahrenheit) for a period 72 hours using a cooling blanket. This treatment appears to protect the brain, decreasing the rate of death and disability and improving the chances of survival and neurodevelopmental outcomes at 18 months correct age. But additional trials are needed to help define the most effective cooling strategies.

The Optimizing Cooling trial will examine whether cooling for a longer time period and/or to a lower temperature will improve the chance of survival and neurodevelopmental outcomes at 18-22 months corrected age. Eligible infants with HIE will be placed in one of four cooling groups: (1) cooling for 72 hours to 33.5°C; (2) cooling for 120 hours to 33.5°C; (3) cooling for 72 hours to 32.0°C; and (4) cooling for 120 hours to 32.0°C. Infants will be monitored closely and receive the care of the Neonatal Intensive Care Unit (NICU).

Infants enrolled in the study will be placed on a cooling blanket - the same type of blanket children's hospitals use in the NICU, in operating rooms during surgeries, and to cool children with high fevers. Each infant will be cooled according to the study group he or she is assigned to. During cooling, the infant's temperature will be very closely monitored by continuous esophageal (core)temperature readings. This will be done by placing a soft, narrow, flexible plastic tube into the infant's nose and down to just above the stomach. Skin temperatures will also be monitored closely. At the end of the assigned period of cooling, the infant will be slowly re-warmed until a normal core temperature of 36.5 to 37.0°C (97.7 to 98.6°C) is reached.

Infants will be examined at 18-22 months corrected age to assess their neurodevelopmental outcomes.

Secondary Studies include:

A. Using aEEG to 1)predict mortality or moderate to severe disability at 18-22 months in term infants with HIE treated with systemic hypothermia and 2) to record electrical seizure activity to compare rewarming initiated at 72 hours and later rewarming that is initiated at 120 hours.

B. Secondary Study includes determining an association between MRI detectable injury and neurodevelopment at 18-22 months.

ELIGIBILITY:
Inclusion Criteria:

Eligibility will be determined in a stepped process:

1. All infants with a gestational age ≥ 36 weeks will be screened for study entry if they are admitted to the NICU with a diagnosis of fetal acidosis, perinatal asphyxia, neonatal depression or encephalopathy.
2. Infants will be eligible if:

   * They have a pH ≤ 7.0 or a base deficit ≥ 16m mEq/ L on umbilical cord or any postnatal sample within 1 hour of age.
   * If, during this interval, they have a pH between 7.01 and 7.15, a base deficit is between 10 and 15.9 mEq/L, or a blood gas is not available, AND they have an acute perinatal event AND either a 10-minute Apgar score ≤ 5 or assisted ventilation initiated at birth and continued for at least 10 minutes.
3. Once these criteria are met, eligible infants will have a standardized neurological examination performed by a certified physician examiner. Infants will be candidates for the study when encephalopathy or seizures are present. For this study, encephalopathy is defined as the presence of 1 or more signs in 3 of the following 6 categories:

   * Level of consciousness: lethargy, stupor or coma;
   * Spontaneous activity: decreased, absent;
   * Posture: distal flexion, decerebrate;
   * tone: hypotonia, flaccid or hypertonia, rigid;
   * Primitive reflexes: a) suck, weak, absent; b) Moro, incomplete, flaccid;
   * Autonomic nervous system: a) pupils: constricted, unequal, skew deviation or non reactive to light; b) heart rate: bradycardia, variable heart rate or c) respiration: periodic breathing, apnea.

Eligible infants from multiple births will be enrolled in the same arm of the study.

Exclusion Criteria:

* Inability to randomize by 6 hours of age
* Major congenital abnormality
* Major chromosomal abnormality (including Trisomy 21),
* Severe growth restriction (≤ 1800gm birth weight),
* Infant is moribund and will not receive any further aggressive treatment,
* Refusal of consent by parent
* Refusal of consent by attending neonatologist
* Infants with a core temperature < 33.5°C for > 1 hour at the time of screening by the research team would not be eligible for the study.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2010-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seetha Shankaran, MD, Study Chair — Wayne State University; Abbot R Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; William Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Barbara Schmidt, MD, MSc, Principal Investigator — University of Pennsylvania; Carl D'Angio, MD, Principal Investigator — University of Rochester; Uday Devaskar, MD, Principal Investigator — University of California, Los Angeles; Leif Nelin, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Derived] Shankaran S, Laptook AR, Guimaraes C, Murnick J, McDonald SA, Das A, Petrie Huitema CM, Pappas A, Higgins RD, Hintz SR, Zaterka-Baxter KM, Van Meurs KP, Sokol GM, Chalak LF, Colaizy TT, Devaskar U, Tyson JE, Reynolds AM, DeMauro SB, Sanchez PJ, Laughon MM, Carlo WA, Watterberg K, Puopolo KM, Hibbs AM, Hamrick SEG, Cotten CM, Barks J, Poindexter BB, Truog WE, D'Angio CT; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. NICHD Magnetic Resonance Brain Imaging Score in Term Infants With Hypoxic-Ischemic Encephalopathy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2025 Apr 1;179(4):383-395. doi: 10.1001/jamapediatrics.2024.6209. PMID 39960680
- [Derived] Bonifacio SL, Chalak LF, Van Meurs KP, Laptook AR, Shankaran S. Neuroprotection for hypoxic-ischemic encephalopathy: Contributions from the neonatal research network. Semin Perinatol. 2022 Nov;46(7):151639. doi: 10.1016/j.semperi.2022.151639. Epub 2022 Jun 10. PMID 35835616
- [Derived] Shukla VV, Bann CM, Ramani M, Ambalavanan N, Peralta-Carcelen M, Hintz SR, Higgins RD, Natarajan G, Laptook AR, Shankaran S, Carlo WA. Predictive Ability of 10-Minute Apgar Scores for Mortality and Neurodevelopmental Disability. Pediatrics. 2022 Apr 1;149(4):e2021054992. doi: 10.1542/peds.2021-054992. PMID 35296895
- [Derived] Chalak LF, Pappas A, Tan S, Das A, Sanchez PJ, Laptook AR, Van Meurs KP, Shankaran S, Bell EF, Davis AS, Heyne RJ, Pedroza C, Poindexter BB, Schibler K, Tyson JE, Ball MB, Bara R, Grisby C, Sokol GM, D'Angio CT, Hamrick SEG, Dysart KC, Cotten CM, Truog WE, Watterberg KL, Timan CJ, Garg M, Carlo WA, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Association Between Increased Seizures During Rewarming After Hypothermia for Neonatal Hypoxic Ischemic Encephalopathy and Abnormal Neurodevelopmental Outcomes at 2-Year Follow-up: A Nested Multisite Cohort Study. JAMA Neurol. 2021 Dec 1;78(12):1484-1493. doi: 10.1001/jamaneurol.2021.3723. PMID 34882200
- [Derived] Ambalavanan N, Shankaran S, Laptook AR, Carper BA, Das A, Carlo WA, Cotten CM, Duncan AF, Higgins RD; EUNICE KENNEDY SHRIVER NICHD NEONATAL RESEARCH NETWORK. Early Determination of Prognosis in Neonatal Moderate or Severe Hypoxic-Ischemic Encephalopathy. Pediatrics. 2021 Jun;147(6):e2020048678. doi: 10.1542/peds.2020-048678. Epub 2021 May 13. PMID 33986149
- [Derived] Shankaran S, Laptook AR, Pappas A, McDonald SA, Das A, Tyson JE, Poindexter BB, Schibler K, Bell EF, Heyne RJ, Pedroza C, Bara R, Van Meurs KP, Huitema CMP, Grisby C, Devaskar U, Ehrenkranz RA, Harmon HM, Chalak LF, DeMauro SB, Garg M, Hartley-McAndrew ME, Khan AM, Walsh MC, Ambalavanan N, Brumbaugh JE, Watterberg KL, Shepherd EG, Hamrick SEG, Barks J, Cotten CM, Kilbride HW, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Effect of Depth and Duration of Cooling on Death or Disability at Age 18 Months Among Neonates With Hypoxic-Ischemic Encephalopathy: A Randomized Clinical Trial. JAMA. 2017 Jul 4;318(1):57-67. doi: 10.1001/jama.2017.7218. PMID 28672318
- [Derived] Pedroza C, Tyson JE, Das A, Laptook A, Bell EF, Shankaran S; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Advantages of Bayesian monitoring methods in deciding whether and when to stop a clinical trial: an example of a neonatal cooling trial. Trials. 2016 Jul 22;17(1):335. doi: 10.1186/s13063-016-1480-4. PMID 27450203
- [Derived] Shankaran S, Laptook AR, Pappas A, McDonald SA, Das A, Tyson JE, Poindexter BB, Schibler K, Bell EF, Heyne RJ, Pedroza C, Bara R, Van Meurs KP, Grisby C, Huitema CM, Garg M, Ehrenkranz RA, Shepherd EG, Chalak LF, Hamrick SE, Khan AM, Reynolds AM, Laughon MM, Truog WE, Dysart KC, Carlo WA, Walsh MC, Watterberg KL, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Effect of depth and duration of cooling on deaths in the NICU among neonates with hypoxic ischemic encephalopathy: a randomized clinical trial. JAMA. 2014 Dec 24-31;312(24):2629-39. doi: 10.1001/jama.2014.16058. PMID 25536254
- [Derived] Shankaran S. Outcomes of hypoxic-ischemic encephalopathy in neonates treated with hypothermia. Clin Perinatol. 2014 Mar;41(1):149-59. doi: 10.1016/j.clp.2013.10.008. PMID 24524452
- See also: Neonatal Research Network website — http://neonatal.rti.org
- Available data/document: Publication — http://www.ncbi.nlm.nih.gov/pubmed/25536254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1261 infants assessed for eligibility. 897 were excluded for not meeting eligibility criteria (N=747) or not having parental or physician consent (N=150).
Pre-assignment Details: All eligible infants with consent were randomized to one of four treatment arms/groups.
Period: Overall Study
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Started | 95 | 90 | 96 | 83
Died Prior to Discharge | 7 | 13 | 15 | 14
Died After Discharge | 1 | 2 | 3 | 1
Completed | 84 | 69 | 75 | 63
Not Completed | 11 | 21 | 21 | 20
Not completed — Death | 8 | 15 | 18 | 15
Not completed — Lost to Follow-up | 3 | 6 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours | Total
Number analyzed (Participants) | 95 | 90 | 96 | 83 | 364
Age, Continuous [Mean (Standard Deviation); unit: hours] — Age at Randomization Population: Data was missing for one participant.
  hours
    number analyzed (Participants) | 95 | 90 | 95 | 83 | 363
    (all) | 5.1 (1.0) | 4.9 (1.2) | 4.8 (1.1) | 5.0 (1.6) | 4.9 (1.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 52 | 53 | 51 | 56 | 212
  Female | 43 | 37 | 44 | 27 | 151
  Ambiguous | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data was missing for six participants.
  Participants
    Black: number analyzed (Participants) | 95 | 89 | 94 | 80 | 358
    Black | 29 | 28 | 32 | 25 | 114
    White: number analyzed (Participants) | 95 | 89 | 94 | 80 | 358
    White | 60 | 56 | 55 | 48 | 219
    Other: number analyzed (Participants) | 95 | 89 | 94 | 80 | 358
    Other | 6 | 5 | 7 | 7 | 25
Birthweight [Mean (Standard Deviation); unit: grams] — Population: Data was missing for one participant.
  grams
    number analyzed (Participants) | 95 | 90 | 95 | 83 | 363
    (all) | 3230 (528) | 3360 (544) | 3354 (676) | 3511 (615) | 3359 (599)
Level of encephalopathy [Count of Participants; unit: Participants]
  Moderate | 74 | 70 | 78 | 58 | 280
  Severe | 21 | 20 | 18 | 25 | 84

OUTCOME MEASURES:

1. Primary Outcome: Death or Moderate to Severe Disability
Description: Death includes any mortality prior to follow up at 18-22 months. Severe disability was defined by any of the following: a Bayley III cognitive score <70, a GMFCS level of 3-5, blindness or profound hearing loss (inability to understand commands despite amplification). Moderate disability was defined as a Bayley cognitive score of 70-84 and either a GMFCS level of 2, seizure disorder, or a hearing deficit requiring amplification to understand commands.
Time Frame: Birth to 22 months corrected age
Population: Includes all deaths and all infants followed at 18-22 months. Does not include 17 infants lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 92 | 84 | 93 | 78
Participants | 27 | 29 | 32 | 22
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — Generalized Estimating Equations models with log link, adjusted for level of encephalopathy and intra-center correlations; Risk Ratio (RR) = 1.23, 95% CI 2-sided [0.76 to 1.98]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.78 to 1.87]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.53 to 1.35]

2. Secondary Outcome: Death
Description: Death includes any mortality prior to follow up at 18-22 months.
Time Frame: Birth to 22 months corrected age
Population: Includes all deaths and all infants followed at 18-22 months. Does not include 17 infants lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 92 | 84 | 93 | 78
Participants | 8 | 15 | 18 | 15
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.16, 95% CI 2-sided [0.55 to 8.49]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 2.52, 95% CI 2-sided [1.06 to 5.95]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.85, 95% CI 2-sided [0.79 to 4.31]

3. Secondary Outcome: Level of Disability Among Survivors
Description: Among survivors number of normal infants and infants with mild, moderate, and severe disability
  Severe disability was defined by any of the following: a Bayley III cognitive score <70, a GMFCS level of 3-5, blindness or profound hearing loss (inability to understand commands despite amplification). Moderate disability was defined as a Bayley cognitive score of 70-84 and either a GMFCS level of 2, seizure disorder, or a hearing deficit requiring amplification to understand commands. Mild impairment was defined by a cognitive score 70-84, or a cognitive score ≥ 85 and any of the following: presence of a GMFCS level 1 or 2, seizure disorder or hearing loss not requiring amplification. Normal was defined by a cognitive score ≥ 85 in the absence of any neurosensory deficits or seizures after NICU discharge.
Time Frame: Follow up at 18-22 months corrected age
Population: Includes all infants followed at 18-22 months except for 6 infants who could not be distinguished between normal and mild. Does not include 17 infants lost to follow up or 56 deaths
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 81 | 69 | 72 | 63
Participants
  Severe disability | 18 | 11 | 14 | 7
  Moderate disability | 1 | 3 | 0 | 0
  Mild disability | 16 | 15 | 22 | 18
  Normal | 46 | 40 | 36 | 38

4. Secondary Outcome: Withdrawal of Care
Description: Number of infants for whom aggressive care is withdrawn
Time Frame: Birth through hospital discharge, average 22 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 95 | 90 | 96 | 83
Participants | 6 | 12 | 14 | 13

5. Secondary Outcome: Clinical Neonatal Seizures
Description: Documented seizures during hospital course
Time Frame: Through death, discharge, or transfer
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 95 | 90 | 96 | 83
Participants | 50 | 43 | 44 | 40

6. Secondary Outcome: Bayley Cognitive Score
Description: Bayley Scale of Infant Development Composite Cognitive Score. The total composite score is reported, ranging from the lowest score of 55 to the highest score of 145. Lower values specify worse outcome.
Time Frame: Follow up at 18-22 months corrected age
Population: Infants who survived and were followed at 18-22 months
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 78 | 69 | 73 | 63
scores on a scale | 90 [80 to 100] | 90 [75 to 100] | 90 [80 to 100] | 90 [80 to 95]

7. Secondary Outcome: Cerebral Palsy
Time Frame: Follow up at 18-22 months corrected age
Population: Infants who survived and were followed at 18-22 months
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 83 | 69 | 75 | 63
Participants | 15 | 13 | 10 | 8
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.23, 95% CI 2-sided [0.64 to 2.38]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.36 to 1.90]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.26 to 1.57]

8. Secondary Outcome: Level of Disability Among Survivors, by Level of HIE
Description: Among survivors, number of normal infants and infants with mild, moderate and severe disability Severe disability was defined by any of the following: a Bayley III cognitive score <70, a GMFCS level of 3-5, blindness or profound hearing loss (inability to understand commands despite amplification). Moderate disability was defined as a Bayley cognitive score of 70-84 and either a GMFCS level of 2, seizure disorder, or a hearing deficit requiring amplification to understand commands. Mild impairment was defined by a cognitive score 70-84, or a cognitive score ≥ 85 and any of the following: presence of a GMFCS level 1 or 2, seizure disorder or hearing loss not requiring amplification. Normal was defined by a cognitive score ≥ 85 in the absence of any neurosensory deficits or seizures after NICU discharge.
Time Frame: Follow up at 18-22 months corrected age
Population: Includes all infants followed at 18-22 months, except for 6 infants who could not be distinguished between normal and mild. Does not include 17 infants lost to follow up or 56 deaths.
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 81 | 69 | 72 | 63
Participants
  Moderate HIE: number analyzed (Participants) | 64 | 60 | 65 | 49
  Moderate HIE: Normal | 41 | 39 | 34 | 31
  Moderate HIE: Mild disability | 13 | 12 | 19 | 13
  Moderate HIE: Moderate disability | 1 | 2 | 0 | 0
  Moderate HIE: Severe disability | 9 | 7 | 12 | 5
  Severe HIE: number analyzed (Participants) | 17 | 9 | 7 | 14
  Severe HIE: Normal | 5 | 1 | 2 | 7
  Severe HIE: Mild disability | 3 | 3 | 3 | 5
  Severe HIE: Moderate disability | 0 | 1 | 0 | 0
  Severe HIE: Severe disability | 9 | 4 | 2 | 2

9. Secondary Outcome: Visual Impairment
Description: Visual impairment is defined as bilateral blindness with some/no useful vision
Time Frame: Follow up at 18-22 months corrected age
Population: Infants who survived and were followed at 18-22 months
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 83 | 69 | 75 | 63
Participants | 6 | 6 | 2 | 4
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.33, 95% CI 2-sided [0.63 to 2.77]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.42, 95% CI 2-sided [0.09 to 2.04]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.20 to 2.99]

10. Secondary Outcome: Hearing Impairment
Description: Hearing impairment is defined as hearing impairment despite amplification
Time Frame: Follow up at 18-22 months corrected age
Population: Infants who survived and were followed at 18-22 months
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 83 | 69 | 75 | 63
Participants | 4 | 2 | 4 | 1
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.14 to 3.01]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 1.31, 95% CI 2-sided [0.44 to 3.91]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.28, 95% CI 2-sided [0.03 to 2.89]

11. Secondary Outcome: Multiple Disabilities
Description: Multiple disabilities is defined as two or more of the following 5 components: disabling CP, GMFCS level 3-5, Bayley cognitive score < 70, blindness, or deafness.
Time Frame: Follow up at 18-22 months corrected age
Population: Infants who survived and were followed at 18-22 months
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 84 | 69 | 75 | 63
Participants | 14 | 9 | 7 | 5
Statistical Analysis 1: Comparison: 33.5°C for 72 Hours vs 32.0°C for 72 Hours; 32.0°C for 72 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.37 to 2.07]
Statistical Analysis 2: Comparison: 33.5°C for 72 Hours vs 33.5°C for 120 Hours; 33.5°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.30 to 1.35]
Statistical Analysis 3: Comparison: 33.5°C for 72 Hours vs 32.0°C for 120 Hours; 32.0°C for 120 hours vs. 33.5°C for 72 hours (33.5°C for 72 hours is the comparison group); Test type: Superiority — [test comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.13 to 1.64]

12. Secondary Outcome: Multiorgan Dysfunction
Description: The data needed for this analysis are not collected directly, and will not be analyzed as the study was terminated early and no funds available to complete this complex analysis. The data for this study will be stored at the NICHD-DASH for investigators.
Time Frame: Until death, discharge, or transfer
Population: No patients were analyzed for this outcome as the study was terminated early and no additional funds available to complete this complex analysis.
Arm/Group | 33.5°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 72 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Severe Neonatal Brain Abnormalities
Description: Total hemispheric devastation based on MRI taken between 7-14 days of life
Time Frame: 7-14 days of life
Population: Note that 66 infants are not included (total N for OC study=364); 49 were excluded due to lack of MRI of adequate quality, 16 due to missing primary outcome, and 1 due to genetic abnormality.
Measure: Count of Participants; unit: Participants
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
Number analyzed (Participants) | 82 | 75 | 80 | 61
Participants
  Total hemispheric devastation = YES | 10 | 11 | 4 | 7
  Total hemispheric devastation = NO | 72 | 64 | 76 | 54

ADVERSE EVENTS:
Time Frame: During study intervention period: 72 or 120 hours from baseline, based on treatment arm
Description: 17 infants lost to follow up were excluded from the All-Cause Mortality table. Mortality cannot be assessed for infants lost to follow up.
Arm/Group | 33.5°C for 72 Hours | 32.0°C for 72 Hours | 33.5°C for 120 Hours | 32.0°C for 120 Hours
All-Cause Mortality (participants affected / at risk) | 8/92 | 15/84 | 18/93 | 15/78
Serious Adverse Events (participants affected / at risk) | 10/95 | 15/90 | 11/96 | 23/83
Other Adverse Events (participants affected / at risk) | 5/95 | 3/90 | 6/96 | 9/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 33.5°C for 72 Hours (N=95) | 32.0°C for 72 Hours (N=90) | 33.5°C for 120 Hours (N=96) | 32.0°C for 120 Hours (N=83)
Death during intervention (Nervous system disorders) | 5 (5) | 5 (5) | 7 (7) | 12 (12)
Cardiac Arrythmia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 7 (9)
Thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major Bleeding (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Other (General disorders) | 5 (7) | 10 (10) | 6 (7) | 11 (16) — Other Serious Adverse Events
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 33.5°C for 72 Hours (N=95) | 32.0°C for 72 Hours (N=90) | 33.5°C for 120 Hours (N=96) | 32.0°C for 120 Hours (N=83)
Metabolic acidosis developing >3 hours after initiation of intervention and persisting >3 hours (General disorders) | 2 (3) | 0 (0) | 1 (1) | 4 (4)
Alteration of Skin Integrity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 5 (8) | 5 (5)

LIMITATIONS AND CAVEATS:
This RCT was stopped for safety and futility reasons by the Data Safety and Monitoring Committee so did not enroll the target number of participants needed to achieve target power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators must adhere to the Neonatal Research Network Publication policies.